CLINICAL TRIAL: NCT05710640
Title: Using the Cholinergic Anti-Inflammatory Pathway to Treat Juvenile Idiopathic Arthritis (AJA01)
Brief Title: Transcutaneous Cervical Vagus Nerve Stimulation (tcVNS) in JIA
Acronym: AJA01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to feasibility concerns and budget constraints.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (ACE) (Unknown); Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT AJA01
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: Juvenile Idiopathic Arthritis; JIA; Children; tcVNS; Cytokines; Inflammation; Nonsignificant risk; NSR
MeSH Terms: conditions — Arthritis, Juvenile; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Blinded phase (Experimental): Participants will receive 5 minutes of active tcVNS or sham tcVNS daily for 8 weeks.
  Interventions: Device: Active tcVNS; Device: Sham tcVNS
- Open-Label phase (Experimental): Participants will receive 5 minutes of stimulation via the active tcVNS device for 8 weeks after a double-blind, sham-controlled 8- week period.
  Interventions: Device: Active tcVNS

INTERVENTIONS:
Device: Active tcVNS — Participants being treated with an active tcVNS device will attach the stimulator, lead, and clip electrode to assemble the complete device and coat the electrode surfaces with electrode gel. The electrode will be placed on the cymba concha of a left ear that is free of earrings or other objects, cleaned internally and externally, and coated with a thin layer of electrode gel. The participant will gradually advance the stimulator knob clockwise until they feel the electrical stimulation at a level that is easily tolerated for 5 minutes and is not painful. The participant will apply the stimulation for 5 minutes, then the participant will turn off the stimulator, remove the electrode from the ear, and clean the ear and electrodes with gauze.
  Other Names: tVNS; Active tVNS; taVNS; Active taVNS
  Arms: Blinded phase
Device: Sham tcVNS — Participants being treated with a sham tcVNS device will place adhesive electrodes on the left side of the neck, which has had neck jewelry removed and has been cleaned at the site of treatment. The participant will then connect the lead to the electrodes and the stimulator to assemble the complete sham tcVNS device. The participant will gradually advance the stimulator knob clockwise until they feel the electrical stimulation at a level that is easily tolerated for 5 minutes and is not painful. Participants in this group will be instructed to not turn the knob above "3" on the dial as this is the maximum acceptable treatment level at the neck. The participant will apply the stimulation for 5 minutes, then the participant will turn off the stimulator, remove the electrode from the neck, and dispose of the electrodes.
  Other Names: tVNS; Sham tVNS; taVNS; Sham taVNS; Sham Stimulation
  Arms: Blinded phase
Device: Active tcVNS — Participants being treated with an active tcVNS device will attach the stimulator, lead, and clip electrode to assemble the complete device and coat the electrode surfaces with electrode gel. The electrode will be placed on the cymba concha of a left ear that is free of earrings or other objects, cleaned internally and externally, and coated with a thin layer of electrode gel. The participant will gradually advance the stimulator knob clockwise until they feel the electrical stimulation at a level that is easily tolerated for 5 minutes and is not painful. The participant will apply the stimulation for 5 minutes, then the participant will turn off the stimulator, remove the electrode from the ear, and clean the ear and electrodes with gauze.
  Other Names: tVNS; Active tVNS; taVNS; Active taVNS
  Arms: Open-Label phase

SUMMARY:
The study is a multicenter, double-blind, sham-controlled trial to evaluate the safety and effectiveness of tcVNS on pain and inflammation associated with JIA. tcVNS is administered with a device that gives off mild electrical impulses through the skin to stimulate the vagus nerve. Part of the vagus nerve and its branches are located in the head and neck. For this study, the impulses will be administered using a small electrode at the cymba concha for participants receiving treatment with active tcVNS and at the neck for participants receiving sham stimulation. The electrode helps to conduct the stimulation through the skin. This stimulation triggers a chemical response through the nerves and has been found to be effective in reducing pain and inflammation in several diseases.

The primary objective of this study is to determine the effect of tcVNS on JIA ACR 50 in participants with active JIA. The components of the active and sham tcVNS devices, utilizing the Roscoe Medical TENS 7000, have been FDA 510(k)-cleared and have been determined by the IRB to be a nonsignificant risk device.

DETAILED DESCRIPTION:
AJA01 is a multicenter, double-blind, sham-controlled, 16-week trial to evaluate the safety and effectiveness of tcVNS for the treatment of JIA.

A total of 100 participants will be randomized 1:1 to treatment with active tcVNS at the cymba concha or sham stimulation at the neck for 5 minutes once a day for 8 weeks. During this time, participants/parents, and participant assessors will be blinded to treatment assignment; treatments on clinic visit days will be conducted in the clinic under the supervision of a trained, unblinded staff member, and participants will only discuss the stimulation procedure with this staff member. An unblinded site investigator will follow up on any safety events. The double-blind, sham-controlled 8-week period will be followed by an 8-week open-label period in which all participants will receive treatment with active tcVNS at the cymba concha once a day for 5 minutes. Participants and their parents will be told it is likely they will feel the stimulation, but it should not be painful.

There are 10 visits for the study, 8 clinic visits and 2 tele-visits. Participants will have physical exams with joint assessments, lab tests, and questionnaire completion by the physicians and participants at each clinic visit. Participants will be trained by the unblinded coordinator to perform stimulation during the clinic visit following the randomization. Participants will perform the stimulation at home for 5 minutes daily. Participants will complete a diary to document the daily stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 5 through 18 years of age (inclusive) at screening.
2. Regarding informed consent and compliance:

   1. If 5 through 6 years of age, the participant's guardian is willing and able to understand and provide informed consent and comply with study protocol.
   2. If 7 through 17 years of age, the participant is willing and able to sign assent and comply with study protocol, and the participant's guardian is willing and able to understand and provide informed consent and comply with study protocol.
   3. If 18 years of age, the participant is willing and able to understand and provide informed consent and comply with study protocol.
3. The participant has a Juvenile Idiopathic Arthritis (JIA) diagnosis meeting International League of Associations for Rheumatology (ILAR) classification criteria with one of the following subtypes:

   1. rheumatoid-factor negative polyarthritis
   2. rheumatoid-factor positive polyarthritis
   3. persistent oligoarthritis
   4. extended oligoarthritis
   5. psoriatic arthritis
   6. enthesitis-related arthritis
   7. systemic arthritis
4. The participant has >=3 joints with active arthritis at screening
5. If the participant is receiving therapy for JIA at screening, that therapy is stable for the time period outlined below and is expected to remain stable for the duration of the study:

   a. stable dose for at least 1 week prior to screening:

   i. Oral steroids, <= 0.2 mg/kg/day with a maximum 10 mg/day dose

   b. stable dose for at least 2 weeks prior to screening:

   i. NSAIDs

   c. stable dose for at least 8 weeks prior to screening:

   i. adalimumab

   ii. anakinra

   iii. canakinumab

   iv. certolizumab pegol

   v. etanercept

   vi. golimumab

   vii. infliximab

   viii. leflunomide

   ix. methotrexate

   x. tocilizumab

   d. stable dose for at least 12 weeks prior to screening:

   i. abatacept
6. If a female of child-bearing potential, the participant has a negative urine pregnancy test at screening
7. If of reproductive potential, must agree to abstinence or effective methods of birth control for the duration of the study

Exclusion Criteria:

1. Other than NSAIDs or intra-articular injections, participant has been treated for JIA with lack of efficacy with:

   1. More than 2 different classes of therapies, or
   2. More than 3 medications in total
2. Participant has received high-dose steroids (>=0.2 mg/kg/day) within the 28 days prior to screening.
3. Participant has had active systemic disease (fever, systemic rash) within the 3 months prior to screening including any of the following lab manifestations at screening:

   1. Ferritin >1000 ng/mL
   2. White blood cell (WBC) ≥15,000/mm^3
4. Participant has had an active acute systemic infection within 2 weeks of screening. involving fever (100.4⁰F or higher) for more than 24 hours, requirement for systemic antibiotics or antivirals, GI symptoms lasting 48 hours or more, or the need to hold second line medications for JIA (methotrexate or biologic).
5. Participant has a history of arrhythmia.
6. Participant has been diagnosed with postural orthostatic tachycardia syndrome (POTS).
7. Participant has received an intra-articular cortisone injection within the 28 days prior to screening.
8. Participant has received treatment with an investigational drug or device during the 28 days prior to screening or within five half-lives of the investigational drug prior to screening/baseline, whichever is the greater length of time.
9. Participant has received chronic treatment with an anti-cholinergic medication, including over the counter medications.
10. Participant has received treatment with rituximab:

    1. Within one year of screening
    2. At any time previously without documented B cell repletion
11. Participant has a comorbid disease that has required treatment with corticosteroids within the past year.
12. Participant has an implantable electronic device such as a pacemaker, defibrillator, hearing aid, cochlear implant, insulin pump or deep brain stimulator.
13. Participant has used cutaneous vagus nerve stimulation within 12 weeks prior to screening.
14. Participant has received a live attenuated viral vaccine within 28 days prior to screening or is expected to receive one during the study.
15. Participant has any condition which, in the opinion of the investigator, would jeopardize the participant's safety following exposure to a study intervention.
16. Participant has any past or current medical problems or findings from a physical examination or laboratory testing that are not listed above but which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or may impact the quality or interpretation of the data obtained from the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Gottlieb, MD, Study Chair — Feinstein Institutes for Medical Research, Cohen Children's Medical Center: Pediatric Rheumatology; Cynthia Aranow, MD, Study Chair — Northwell Health; Timir Datta-Chaudhuri, PhD, Study Chair — Northwell Health; Betty Diamond, MD, Study Chair — Northwell Health
Locations (7):
- United States (7):
  - University of California San Francisco School of Medicine: Department of Pediatrics, Division of Pediatric Rheumatology, San Francisco, California
  - Nemours Children's Health: Department of Pediatric Rheumatology, Orlando, Florida
  - Indiana University Medical Center: Riley Hospital for Children Department of Pediatric Rheumatology, Indianapolis, Indiana
  - Feinstein Institutes for Medical Research, Cohen Children's Medical Center: Pediatric Rheumatology, Lake Success, New York
  - Stephen D. Hassenfield Children's Center at NYU Langone Health, New York, New York
  - Division of Pediatric Rheumatology at the University of Utah School of Medicine and Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital: Rheumatology Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from the Division of Allergy Immunology and Transplantation-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: Autoimmunity Centers of Excellence (ACE) — https://www.autoimmunitycenters.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tcVNS: Participants in the Active tcVNS arm stimulated themselves for 5 minutes daily with the investigational device at the cymba concha through Week 16.
- Sham Stimulation: Participants in the Sham Stimulation arm stimulated themselves for 5 minutes daily with sham stimulation at the neck through the day prior to the Week 8 visit and then stimulated for 5 minutes daily with active tcVNS at the cymba concha using the investigational device from Week 8 through Week 16.
Period: Overall Study
Arm/Group | Active tcVNS | Sham Stimulation
Started | 9 (One participant randomized but did not initiate stimulation.) | 9
Completed | 7 | 8
Not Completed | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrew prior to first device stimulation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat (mITT) population included all randomized participants who received any active tcVNS stimulation or sham stimulation.
Groups:
- Active tcVNS: Participants in the Active tcVNS arm stimulated themselves for 5 minutes daily with the investigation device at the cymba concha through Week 16.
- Total: Total of all reporting groups
Arm/Group | Active tcVNS | Sham Stimulation | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (3.36) | 14.1 (3.37) | 13.6 (3.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 5 | 7 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17
JIA Subtype [Count of Participants; unit: Participants] — JIA subtype at Baseline
  Participants
    Rheumatoid-factor negative polyarthritis | 5 | 6 | 11
    Rheumatoid-factor positive polyarthritis | 1 | 1 | 2
    Persistent oligoarthritis | 1 | 0 | 1
    Extended oligoarthritis | 0 | 1 | 1
    Psoriatic arthritis | 0 | 0 | 0
    Enthesitis-related arthritis | 1 | 1 | 2
    Systemic arthritis | 0 | 0 | 0
Number of Joints with Active Arthritis [Mean (Standard Deviation); unit: Joints] — Number of joints with active arthritis at Baseline. Active arthritis is non-boney swelling (joint effusion) or limitation of motion accompanied by warmth, pain on motion or tenderness to palpation.
  Joints | 9.5 (6.48) | 8.2 (3.60) | 8.8 (5.03)
Number of Joints with Limited Motion [Mean (Standard Deviation); unit: Joints] — Number of joints with limitation of motion at Baseline.
  Joints | 4.1 (6.92) | 4.6 (3.17) | 4.4 (5.10)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 50 Responders at Week 8 Compared to Baseline
Description: The JIA ACR 50 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 50 is achieved if 3 of any 6 core set variables improved by at least 50% from Baseline, and no more than 1 variable worsens by >30%. A negative change from Baseline in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at Week 8 are imputed as JIA ACR 50 non-responders at Week 8.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of Participants | 0.250 [0.032 to 0.651] | 0.333 [0.075 to 0.701]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Test type: Superiority; p = 1.000, Fisher Exact — P-value is from comparing the proportion of JIA ACR 50 Responders between the two device groups using a Fisher's exact test

2. Secondary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 50 Responders at Weeks 4, 12, and 16 Compared to Baseline
Description: The JIA ACR 50 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 50 is achieved if 3 of any 6 core set variables improved by at least 50% from Baseline, and no more than 1 variable worsens by >30%. A negative change from Baseline in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at any visit are imputed as JIA ACR 50 non-responders at that visit.
Time Frame: Weeks 4, 12, 16
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of participants
  Week 4 | 0.375 [0.085 to 0.755] | 0.111 [0.003 to 0.482]
  Week 12 | 0.625 [0.245 to 0.915] | 0.444 [0.137 to 0.788]
  Week 16 | 0.625 [0.245 to 0.915] | 0.556 [0.212 to 0.863]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 4; Test type: Superiority; p = 0.294, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 0.637, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 1.00, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 Responders at Weeks 4, 8, 12, and 16 Compared to Baseline
Description: The JIA ACR 30 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 30 is achieved if 3 of any 6 core set variables improved by at least 30% from Baseline, and no more than 1 variable worsens by >30%. A negative change from Baseline in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at any visit are imputed as JIA ACR 30 non-responders at that visit.
Time Frame: Weeks 4, 8, 12, 16
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of participants
  Week 4 | 0.500 [0.157 to 0.843] | 0.556 [0.212 to 0.863]
  Week 8 | 0.375 [0.085 to 0.755] | 0.444 [0.137 to 0.788]
  Week 12 | 0.750 [0.349 to 0.968] | 0.556 [0.212 to 0.863]
  Week 16 | 0.875 [0.473 to 0.997] | 0.667 [0.299 to 0.925]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 4; Test type: Superiority; p = 1.000, Fisher Exact — P-value is from comparing the proportion of JIA ACR 30 Responders between the two device groups using a Fisher's exact test
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 8; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 0.620, Fisher Exact — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 0.576, Fisher Exact — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 70 Responders at Week 4, 8, 12, and 16 Compared to Baseline
Description: The JIA ACR 70 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 70 is achieved if 3 of any 6 core set variables improved by at least 70% from Baseline, and no more than 1 variable worsens by >30%. A negative change from Baseline in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at any visit are imputed as JIA ACR 70 non-responders at that visit.
Time Frame: Weeks 4, 8, 12, 16
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of participants
  Week 4 | 0.125 [0.003 to 0.527] | 0.111 [0.003 to 0.482]
  Week 8 | 0.125 [0.003 to 0.527] | 0.111 [0.003 to 0.482]
  Week 12 | 0.250 [0.032 to 0.651] | 0.333 [0.075 to 0.701]
  Week 16 | 0.500 [0.157 to 0.843] | 0.333 [0.075 to 0.701]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 4; Test type: Superiority; p = 1.000, Fisher Exact — P-value is from comparing the proportion of JIA ACR 70 Responders between the two device groups using a Fisher's exact test
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 8; Test type: Superiority; p = 1.00, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 0.637, Fisher Exact — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Juvenile Arthritis Disease Activity Score in 27 Joints (JADAS-27) at Weeks 4, 8, 12, and 16
Description: The JADAS-27 is a measurement of disease activity and is determined by adding the scores of its 4 components: physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); number of joints with active arthritis; and a laboratory measure of inflammation, c-Reactive Protein (CRP), normalized to a value between 0 and 10. The JADAS-27 includes the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), proximal inter-phalangeal joints, hips, knees, and ankles. This provides a score in the range of 0-57 with higher scores indicating worse disease activity. A negative change from Baseline signifies improvement.
Time Frame: Baseline; Weeks 4, 8, 12, 16
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Score on a scale
  Week 4: number analyzed (Participants) | 7 | 9
  Week 4 | -5.187 [-9.741 to -0.633] | -2.350 [-6.366 to 1.666]
  Week 8: number analyzed (Participants) | 7 | 9
  Week 8 | -5.463 [-9.624 to -1.303] | -3.657 [-7.312 to -0.003]
  Week 12: number analyzed (Participants) | 7 | 8
  Week 12 | -9.647 [-12.525 to -6.768] | -7.607 [-10.297 to -4.917]
  Week 16: number analyzed (Participants) | 7 | 8
  Week 16 | -9.722 [-13.267 to -6.178] | -6.256 [-9.568 to -2.943]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 4; Test type: Superiority; p = 0.331, ANCOVA — P-value comes from an analysis of covariance with an outcome of change in JADAS-27 from Baseline and covariates of treatment and Baseline JADAS-27 score
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 8; Test type: Superiority; p = 0.500, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 0.285, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 0.148, ANCOVA — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 50 Responders at Weeks 12 and 16 Compared to Week 8
Description: The JIA ACR 50 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 50 is achieved if 3 of any 6 core set variables improved by at least 50% from Week 8, and no more than 1 variable worsens by >30%. A negative change from Week 8 in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at any visit are imputed as JIA ACR 50 non-responders at that visit.
Time Frame: Week 12 and 16
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of Participants
  Week 12 | 0.125 [0.003 to 0.527] | 0.444 [0.137 to 0.788]
  Week 16 | 0.250 [0.032 to 0.651] | 0.333 [0.075 to 0.701]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 0.294, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 Responders at Weeks 12 and 16 Compared to Week 8
Description: The JIA ACR 30 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 30 is achieved if 3 of any 6 core set variables improved by at least 30% from Week 8, and no more than 1 variable worsens by >30%. A negative change from Week 8 in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at any visit are imputed as JIA ACR 30 non-responders at that visit.
Time Frame: At Weeks 12 and 16
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of Participants
  Week 12 | 0.250 [0.032 to 0.651] | 0.556 [0.212 to 0.863]
  Week 16 | 0.375 [0.085 to 0.755] | 0.333 [0.075 to 0.701]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 0.335, Fisher Exact — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority — P-value is from comparing the proportion of JIA ACR 30 Responders between the two device groups using a Fisher's exact test; p = 1.000, Fisher Exact

8. Secondary Outcome: Proportion of Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 70 Responders at Week 12 and 16 Compared to Week 8
Description: The JIA ACR 70 is a validated composite response consisting of 6 core criteria: number of joints with active arthritis; number of joints with limited motion; physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); a validated measure of physical function, Childhood Health Assessment Questionnaire (CHAQ); and a laboratory measure of inflammation, c-Reactive Protein (CRP). The JIA ACR 70 is achieved if 3 of any 6 core set variables improved by at least 70% from Week 8, and no more than 1 variable worsens by >30%. A negative change from Week 8 in any of the core set variables signifies improvement. Participants missing any of the JIA ACR core criteria at any visit are imputed as JIA ACR 70 non-responders at that visit.
Time Frame: Weeks 12 and 16
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Proportion of Participants
  Week 12 | 0.000 [0.000 to 0.369] | 0.111 [0.003 to 0.482]
  Week 16 | 0.000 [0.000 to 0.369] | 0.222 [0.028 to 0.600]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 0.471, Fisher Exact — [p-value comment as in outcome 4, analysis 1]

9. Secondary Outcome: Change From Week 8 in Juvenile Arthritis Disease Activity Score in 27 Joints (JADAS-27)
Description: The JADAS-27 is a measurement of disease activity and is determined by adding the scores of its 4 components: physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); number of joints with active arthritis; and a laboratory measure of inflammation, c-Reactive Protein (CRP) normalized to a value between 0-10. The JADAS-27 includes the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), proximal inter-phalangeal joints, hips, knees, and ankles. This provides a score in the range of 0-57 with higher scores indicating worse disease activity. A negative change from Week 8 signifies improvement.
Time Frame: Weeks 12 and 16
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Score on a scale
  Week 12: number analyzed (Participants) | 7 | 8
  Week 12 | -5.216 [-7.705 to -2.728] | -4.334 [-6.653 to -2.015]
  Week 16: number analyzed (Participants) | 7 | 8
  Week 16 | -5.211 [-8.559 to -1.863] | -3.053 [-6.173 to 0.068]
Statistical Analysis 1: Comparison: Active tcVNS vs Sham Stimulation; Week 12; Test type: Superiority; p = 0.592, ANCOVA — P-value comes from an analysis of covariance with an outcome of change in JADAS-27 from Week 8 and covariates of treatment and Week 8 JADAS-27 score
Statistical Analysis 2: Comparison: Active tcVNS vs Sham Stimulation; Week 16; Test type: Superiority; p = 0.337, ANCOVA — [p-value comment as in outcome 9, analysis 1]

10. Secondary Outcome: Longitudinal Trends From Baseline to Week 16 in Juvenile Arthritis Disease Activity Score in 27 Joints (JADAS-27)
Description: The JADAS-27 is a measurement of disease activity and is determined by adding the scores of its 4 components: physician's assessment of disease activity (measured on a 10 cm visual analogue scale (VAS)); parent/patient assessment of overall well-being (measured on a 10 cm VAS); number of joints with active arthritis; and a laboratory measure of inflammation, c-Reactive Protein (CRP) normalized to a value between 0-10. The JADAS-27 includes the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), proximal inter-phalangeal joints, hips, knees, and ankles. This provides a score in the range of 0-57 with higher scores indicating worse disease activity.
Time Frame: Baseline; Weeks 4, 8, 12, 16
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Active tcVNS | Sham Stimulation
Number analyzed (Participants) | 8 | 9
Score on a scale
  Baseline | 16.200 (2.5385) | 15.729 (1.6774)
  Week 4: number analyzed (Participants) | 7 | 9
  Week 4 | 10.957 (2.7589) | 13.445 (2.2339)
  Week 8: number analyzed (Participants) | 7 | 9
  Week 8 | 8.686 (1.8442) | 11.767 (1.9662)
  Week 12: number analyzed (Participants) | 7 | 8
  Week 12 | 4.331 (0.8174) | 7.150 (1.8689)
  Week 16: number analyzed (Participants) | 7 | 8
  Week 16 | 4.100 (1.0433) | 8.638 (2.4012)

11. Secondary Outcome: Number of Participants With a Treatment-emergent Adverse Event From Day 0 to Week 8.
Description: A participant who experienced any of the following untoward or unfavorable medical occurrence(s) associated with the investigational device or any study mandated procedures following the first stimulation on Day 0 and prior to the Week 8 visit:
  * Grade 1 or higher mild palpitations, documented arrhythmia, or any unpleasant sensations caused by palpitations
  * Grade 1 or higher stimulation site reactions such as cutaneous irritation, pain, or skin burns
  * Grade 1 or higher Ear and labyrinth disorders as listed in the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, except those of the middle ear
  * Grade 1 or higher JIA flares
  * All other Grade 2 and higher AEs
Time Frame: Day 0 to Week 8
Population: The Blinded Phase Safety population included all participants who received any active tcVNS stimulation or sham stimulation from Day 0 through the day before the Week 8 visit.
Measure: Count of Participants; unit: Participants
Groups:
- Blinded Phase: Active tcVNS: Participants stimulated themselves for 5 minutes daily with active tcVNS at the cymba concha using the investigational device through the day prior to the Week 8 visit.
- Blinded Phase: Sham Stimulation: Participants stimulated themselves for 5 minutes daily with sham stimulation at the neck through the day prior to the Week 8 visit.
Arm/Group | Blinded Phase: Active tcVNS | Blinded Phase: Sham Stimulation
Number analyzed (Participants) | 8 | 9
Participants | 3 | 0

12. Secondary Outcome: Number of Participants With a Treatment-emergent Adverse Event From Week 8 to Week 16
Description: A participant who experienced any of the following untoward or unfavorable medical occurrence(s) associated with the investigational device or any study mandated procedures between Week 8 and Week 16:
  * Grade 1 or higher mild palpitations, documented arrhythmia, or any unpleasant sensations caused by palpitations
  * Grade 1 or higher stimulation site reactions such as cutaneous irritation, pain, or skin burns
  * Grade 1 or higher Ear and labyrinth disorders as listed in the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, except those of the middle ear
  * Grade 1 or higher JIA flares
  * All other Grade 2 and higher AEs
Time Frame: Week 8 to Week 16
Population: The Open-Label Phase Safety population included all participants who received any active tcVNS stimulation on or after the Week 8 visit.
Measure: Count of Participants; unit: Participants
Groups:
- Open-Label Phase: Active tcVNS Following Active tcVNS: Participants stimulated themselves for 5 minutes daily with active tcVNS using the investigational device at the cymba concha from Week 8 through Week 16, following active tcVNS in the 8-week blinded period. Participants are only included in the Open-Label Phase if they stimulated at least once on or after the Week 8 visit.
- Open-Label Phase: Active tcVNS Following Sham Stimulation: Participants stimulated themselves for 5 minutes daily with active tcVNS at the cymba concha using the investigational device from Week 8 through Week 16, following sham stimulation in the 8-week blinded period. Participants are only included in the Open-Label Phase if they stimulated at least once on or after the Week 8 visit.
Arm/Group | Open-Label Phase: Active tcVNS Following Active tcVNS | Open-Label Phase: Active tcVNS Following Sham Stimulation
Number analyzed (Participants) | 7 | 8
Participants | 2 | 1

13. Secondary Outcome: Number of Participants With a Treatment-emergent Serious Adverse Event From Day 0 to Week 8
Description: A participant who experienced any serious untoward or unfavorable medical occurrence(s) associated with the investigational device or any study mandated procedures following the first stimulation on Day 0 and prior to the Week 8 visit.
Time Frame: Day 0 to Week 8
Population: The Blinded Phase Safety population included all participants who received any active tcVNS stimulation or sham stimulation from Day 0 to the day before the Week 8 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Phase: Active tcVNS | Blinded Phase: Sham Stimulation
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With a Treatment-emergent Serious Adverse Event From Week 8 to Week 16
Description: A participant who experienced any serious untoward or unfavorable medical occurrence(s) associated with the investigational device or any study mandated procedures between Week 8 and Week 16.
Time Frame: Week 8 to Week 16
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Phase: Active tcVNS Following Active tcVNS | Open-Label Phase: Active tcVNS Following Sham Stimulation
Number analyzed (Participants) | 7 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were recorded in EDC from after initiation of stimulation at Day 0 to Week 16.
Description: The following AEs were recorded in EDC:
  * Grade 1 or higher mild palpitations, documented arrhythmia, or any unpleasant sensations caused by palpitations
  * Grade 1 or higher stimulation site reactions such as cutaneous irritation, pain, or skin burns
  * Grade 1 or higher Ear and labyrinth disorders as listed in the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, except those of the middle ear
  * Grade 1 or higher JIA flares
  * All other Grade 2 and higher AEs
Arm/Group | Blinded Phase: Active tcVNS | Blinded Phase: Sham Stimulation | Open-Label Phase: Active tcVNS Following Active tcVNS | Open-Label Phase: Active tcVNS Following Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 0/9 | 2/7 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Phase: Active tcVNS (N=8) | Blinded Phase: Sham Stimulation (N=9) | Open-Label Phase: Active tcVNS Following Active tcVNS (N=7) | Open-Label Phase: Active tcVNS Following Sham Stimulation (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT05710640/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT05710640/ICF_000.pdf